CLINICAL TRIAL: NCT02093091
Title: Two-year Clinical Performance in Primary Teeth of Nano-filled Versus Conventional Resin Modified Glass Ionomer Restorations
Brief Title: Clinical Evaluation of Nanoionomer Filling in Primary Teeth
Acronym: CENFPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dr. Sahar E. Abo-Hamar, Doctor (DMD, PhD), Tanta University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TantaU-Nano
Record Dates: First submitted 2014-03-11; First posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Dental Caries
Keywords: nano-filled resin modified glass ionomer; clinical performance; class I; primary teeth; dentin bond strength; Filling of class I
MeSH Terms: conditions — Dental Caries | interventions — Ketac Nano

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitremer (Sham Comparator): Dental caries was removed from primary molars and was filled with the conventional filling material;Vitremer (n = 30). The right molars was always filled by Vitremer. A split-mouth design was used in the present clinical trial. Twenty nine children were involved in the present study and every one had one bilateral identical pair of carious molars except one child that had two identical pairs. This design was performed to enhance the accuracy of the present study.
  Interventions: Procedure: Dental caries was removed from primary molars and was filled with the conventional filling material;Vitremer
- Ketac Nano (Active Comparator): Dental caries was removed from primary molars and was filled with the recent filling material; Ketac Nano (n=30). The left molars was always restored with Ketac Nano filling material.
  Interventions: Procedure: Dental caries was removed from primary molars and was filled with the recent filling material; Ketac Nano.

INTERVENTIONS:
Procedure: Dental caries was removed from primary molars and was filled with the recent filling material; Ketac Nano. — Class I carious primary molars were selected. Dental caries was removed and cavities were prepared. The recent nano-filled RMGI filling (Ketac Nano) was used to fill these cavities.
  Arms: Ketac Nano
Procedure: Dental caries was removed from primary molars and was filled with the conventional filling material;Vitremer — Class I carious primary molars were selected. Dental caries was removed and cavities were prepared. The conventional RMGI filling (Vitremer) was used to fill these cavities.
  Arms: Vitremer

SUMMARY:
This clinical trial was performed to evaluate the nano-filled resin modified glass ionomer (RMGI) -with a brand name of "Ketac Nano"- as a filling material for the treatment of caries in primary teeth. Children aged 5-8 years were selected and treated with either Ketac Nano or another conventional RMGI called Vitremer. Then, the treated children were evaluated at baseline, after one yeat and after two years. The hypothesis to be tested in the present study was: The clinical performance of nano-filled RMGI (Ketac Nano) in class I primary molars will differ from that of its preceding conventional RMGI (Vitremer).

DETAILED DESCRIPTION:
First, shear bond strength of each material to primary molars dentin specimens were measured (n=10) using a notched-edge crosshead. Independent sample t-test was used for statistical analysis. Then, a split mouth designed clinical trial was performed in which nano-filled RMGI; Ketac Nano (KN) and conventional RMGI; Vitremer (VR) were used to restore class I cavities of primary molars. Each material group (n=30) was evaluated according to the modified United States Public Health Service (USPHS) regarding marginal discoloration, marginal adaptation, color match, anatomic form and recurrent caries, at baseline, after one year and after two years. Wilcoxon signed- rank test and Chi-square test were used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* The presence of a bilateral identical pair of primary molars in the same arch containing initial occlusal caries (a minimum of two pits or fissures without any cusp destruction).

Exclusion Criteria:

* Handicapped or uncooperative children and children with extensive or rampant caries.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Evidence of clinically definite deterioration of the evaluated filling materials at specific characters (parameters); marginal discoloration, marginal adaptation, color match, anatomic form and recurrent caries. | 2 years
  The filling materials were blindly evaluated by two trained investigators at specific characters or parameters according to the modified United States Public Health Service (USPHS). Each parameter has three grades of evaluation; Alfa (A), Bravo (B) and Charlie (C) that represent the degree of deterioration of the filling materials.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar E. Abo-Hamar, DMD, PhD, Principal Investigator — Tanta University, Faculty of Dentistry
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt